CLINICAL TRIAL: NCT03357653
Title: A Randomized, Double Blinded, Placebo-controlled, Multicenter, Phase III Study to Evaluate the Efficacy and Safety of Losartan in Early Immunoglobulin A Nephropathy (IgAN) Patients
Brief Title: Beginning of Effective and Safe Treatment in Immunoglobulin A-1 Nephropathy-1
Acronym: BEST-IgAN-1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ewha Womans University (Other)
Collaborators: The Catholic University of Korea (Other); Kyung Hee University Hospital at Gangdong (Other); Kyungpook National University Hospital (Other); Korea University Guro Hospital (Other); SMG-SNU Boramae Medical Center (Other); Seoul National University Bundang Hospital (Other); Seoul National University Hospital (Other); Ajou University School of Medicine (Other); Pusan National University Yangsan Hospital (Other); Severance Hospital (Other); Eulji General Hospital (Other); National Health Insurance Service Ilsan Hospital (Other); Chonnam National University Hospital (Other); Chonbuk National University Hospital (Other); Kangdong Sacred Heart Hospital (Other); Hallym University Medical Center (Other); Gangnam Severance Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BEST-IGAN-001
Record Dates: First submitted 2017-11-15; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Glomerulonephritis, Immunoglobulin A (IgA)
Keywords: proteinuria; progression; early immunoglobulin A (IgA) nephropathy
MeSH Terms: conditions — Glomerulonephritis; Proteinuria; Disease Progression; Kidney Diseases | interventions — Losartan

STUDY DESIGN:
Intervention Model Description: The investigators will test the effect of ARB to prevent the development of significant proteinuria, defined as random urine protein-to-creatinine ratio of >1g/g creatinine. In this study, the investigators choose losartan as a testing ARB. The investigators will compare the rate of significant proteinuria development between 2 arms, namely losartan group and placebo group after 144 weeks' treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan group (Experimental): Losartan 50 mg daily
  Interventions: Drug: Losartan group
- Placebo group (Placebo Comparator): Placebo 1 pill daily which has same size, color and taste with losartan
  Interventions: Drug: Placebo group

INTERVENTIONS:
Drug: Losartan group — Losartan 50 mg daily
  Other Names: Losartan
  Arms: Losartan group
Drug: Placebo group — Placebo 1 pill daily
  Other Names: Placebo
  Arms: Placebo group

SUMMARY:
Immunoglobulin A nephropathy (IgAN) is the most common glomerulonephritis worldwide. IgAN is progressive, particularly when patients have a significant proteinuria (proteinuria >1g/g creatinine), impaired kidney function, or elevated blood pressure. In 10 years, nearly 20-40% of these IgAN patients progress to end-stage renal disease (ESRD). Early IgAN is tentatively defined when proteinuria is insignificant and kidney function and blood pressure are normal. Patients with early IgAN rarely progress to ESRD. However, 30-40% of patients with early IgAN ultimately developed a significant proteinuria and hypertension in 10 years. Therefore, earlier intervention may be needed if it can prevent the development of a significant proteinuria and hypertension. Since angiotensin ll receptor blocker (ARB) is drug of choice in reducing proteinuria and controlling blood pressure, the investigators hypothesized that early introduction of ARB may be beneficial in preventing the significant proteinuria development in early IgAN patients. To prove the hypothesis, the investigators plan the current interventional study.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven IgAN: dominant or co-dominant deposits of mesangial IgA in immunofluorescence stain
2. Age >= 19 years
3. Random urine protein-to-creatinine ratio 0.3 g/g creatinine to 1.0 g/g creatinine at visit 1
4. Estimated glomerular filtration rate >= 60 mL/min/1.73m2 at visit 1
5. People who voluntarily agreed to participate
6. People who are compliant

Exclusion Criteria:

1. Prevalent Hypertension: systolic blood pressure >=140 mmHg and >=90 mmHg, previous physician diagnosis of hypertension, or taking anti-hypertensive drugs
2. Prevalent Diabetes: fasting glucose >= 126 mg/dL, HbA1c >= 6.5%, taking insulin or anti-diabetic drugs, or previous physician diagnosis of diabetes
3. Previous immunosuppressive drugs use to treat IgAN
4. Secondary IgAN
5. Renin-angiotensin-aldosterone inhibitors (RASI) dependent patients (congestive heart failure, ischemic heart disease, and others)
6. hypersensitivity to RASI
7. Other chronic diseases: malignancy within 5 years, significant liver and gastrointestinal disease and other autoimmune disease
8. Pregnancy
9. symptomatic orthostatic hypotension
10. People who already participated in other interventional studies or taking interventional drugs within 3 month of screening visit
11. Inappropriate people ascertained by investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2018-01-30 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Significant proteinuria rate | 144 weeks after study started
  Random urine protein-to-creatinine ratio >= 1g/g creatinine

SECONDARY OUTCOMES:
Proteinuria remission rate | 48 weeks, 96 weeks, and 144 weeks after study started
  Random urine protein-to-creatinine ratio < 0.20 g/g creatinine
Impaired kidney function rate | 48 weeks, 96 weeks, and 144 weeks after study started
  estimated glomerular filtration rate decline >= 40% from the baseline value
Hypertension development rate | 48 weeks, 96 weeks, and 144 weeks after study started
  Systolic blood pressure >= 140 or diastolic blood pressure >= 90

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ryeol Ryu, Professor, Principal Investigator — Ewha Womans University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li PK, Kwan BC, Chow KM, Leung CB, Szeto CC. Treatment of early immunoglobulin A nephropathy by angiotensin-converting enzyme inhibitor. Am J Med. 2013 Feb;126(2):162-8. doi: 10.1016/j.amjmed.2012.06.028. PMID 23331443
- [Background] Jo YI, Na HY, Moon JY, Han SW, Yang DH, Lee SH, Park HC, Choi HY, Lim SD, Kie JH, Lee YK, Shin SK. Effect of low-dose valsartan on proteinuria in normotensive immunoglobulin A nephropathy with minimal proteinuria: a randomized trial. Korean J Intern Med. 2016 Mar;31(2):335-43. doi: 10.3904/kjim.2014.266. Epub 2016 Feb 15. PMID 26874511
- [Background] Nieuwhof C, Kruytzer M, Frederiks P, van Breda Vriesman PJ. Chronicity index and mesangial IgG deposition are risk factors for hypertension and renal failure in early IgA nephropathy. Am J Kidney Dis. 1998 Jun;31(6):962-70. doi: 10.1053/ajkd.1998.v31.pm9631840.
- [Background] Lai FM, Szeto CC, Choi PC, Li PK, Chan AW, Tang NL, Lui SF, Wang AY, To KF. Characterization of early IgA nephropathy. Am J Kidney Dis. 2000 Oct;36(4):703-8. doi: 10.1053/ajkd.2000.17614. PMID 11007671
- [Background] Szeto CC, Lai FM, To KF, Wong TY, Chow KM, Choi PC, Lui SF, Li PK. The natural history of immunoglobulin a nephropathy among patients with hematuria and minimal proteinuria. Am J Med. 2001 Apr 15;110(6):434-7. doi: 10.1016/s0002-9343(01)00659-3. PMID 11331053
- [Background] Shen P, He L, Li Y, Wang Y, Chan M. Natural history and prognostic factors of IgA nephropathy presented with isolated microscopic hematuria in Chinese patients. Nephron Clin Pract. 2007;106(4):c157-61. doi: 10.1159/000104426. Epub 2007 Jun 26. PMID 17596724
- [Background] Lee H, Hwang JH, Paik JH, Ryu HJ, Kim DK, Chin HJ, Oh YK, Joo KW, Lim CS, Kim YS, Lee JP. Long-term prognosis of clinically early IgA nephropathy is not always favorable. BMC Nephrol. 2014 Jun 19;15:94. doi: 10.1186/1471-2369-15-94. PMID 24946688
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT03357653/Prot_SAP_000.pdf